CLINICAL TRIAL: NCT02381405
Title: A Randomized Open Label Study Evaluating a Proprietary Amino Acid Mixture (Enterade®)- for Maintaining Bowel Regularity in Patients With GI Toxicity From Any Combination of Therapy Including Tyrosine Kinase Inhibitors (TKI)
Brief Title: A Study Evaluating a Proprietary Amino Acid Mixture (Enterade®)- for Maintaining Bowel Regularity in Patients With GI Toxicity From Any Combination of Therapy Including Tyrosine Kinase Inhibitors (TKI)
Status: Terminated | Phase: Not Applicable | Type: Interventional
Sponsor: GenesisCare USA (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Enterade 11/11/14
Record Dates: First submitted 2015-03-03; First posted 2015-03-06 (Estimated); Last update posted 2020-01-13 (Actual); Status verified 2020-01

CONDITIONS: Diarrhea
MeSH Terms: conditions — Diarrhea

ARMS (2):
- A (Active Comparator): Enterade beverage
  Interventions: Dietary Supplement: Enterade beverage
- B (No Intervention): Standard of care

INTERVENTIONS:
Dietary Supplement: Enterade beverage
  Arms: A

SUMMARY:
This is an open label, randomized investigation of a proprietary blend of amino acids, called Enterade®, and its effect on irregularity (diarrhea) caused by radiation therapy and/or chemotherapy including TKI*. Subjects will be randomized to receive Enterade® or continue standard of care. Two patients will be enrolled on the treatment arm for each patient on the control arm.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with any combination of therapies including radiation therapy alone, chemotherapy alone, TKI alone, or any combination are eligible.
2. This includes patients with therapies including Xeloda (capecitabine), Camptosar (irinotecan) or 5-FU (fluorouracil) with cancer.
3. Patients who have been diagnosed with a CID CTCAE toxicity of grade 3 or higher
4. Patients must be at least 18 years of age.
5. ECOG performance status 0-2.
6. Patients must have diarrhea symptoms, judged secondary to the systemic therapy, combined systemic therapy, and/or radiation, and must be requiring loperamide or similar (Imodium®) for symptom management. For the purposes of this study, diarrhea will be defined as three or more loose or liquid stools per day or loose watery stool (greater volume of stool) that occur more frequently than usual and lasting for more than three days.

Exclusion Criteria:

1. ECOG performance status 3 or greater.
2. Pregnant and/or breast-feeding women
3. Pre-menopausal subjects as well as subjects with ovarian radiation or concomitant treatment with an LH-RH agonist/antagonist must have a negative pregnancy test and agree to use an adequate method of contraception as recommended by their treating physicians
4. Post-menopausal status is defined either by:

   1. age ≥55 years and one year or more of amenorrhea,
   2. age <55 years and one year or more of amenorrhea with an estradiol assay <20 pg/mL
   3. bilateral oophorectomy
   4. CID CTCAE grade 1 or 2 (not requiring Loperamide or similar)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2015-02; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Patient reported gastrointestinal (GI) symptoms using EPIC | 12 Days

CONTACTS AND LOCATIONS:
Locations (1):
- 21st Century Oncology, Jacksonville, Florida, United States